CLINICAL TRIAL: NCT01176968
Title: A Double-blind, Randomized, Placebo-controlled Trial Evaluating The Safety And Efficacy Of Early Treatment With Eplerenone In Patients With Acute Myocardial Infarction
Brief Title: Impact Of Eplerenone On Cardiovascular Outcomes In Patients Post Myocardial Infarction
Acronym: REMINDER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A6141116; 2010-019844-38 (EudraCT Number); REMINDER (Other: Alias Study Number)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction
Keywords: Eplerenone; myocardial infarction; mortality; morbidity
MeSH Terms: conditions — Myocardial Infarction | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone plus standard of care (Experimental)
  Interventions: Drug: Eplerenone
- Placebo plus standard of care (Placebo Comparator): Matching placebo for eplerenone 25mg film coated tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — Maximum dose of 2x25 mg film coated tablets per day for the duration of the study (approximately 18 months maximum). Lower doses may be administered determined by blood biochemistry data.
  Other Names: Inspra
  Arms: Eplerenone plus standard of care
Drug: Placebo — Matching placebo tablets
  Arms: Placebo plus standard of care

SUMMARY:
Administration of eplerenone within 24 hours of onset of symptoms of myocardial infarction, in patients without heart failure, reduces cardiovascular mortality / morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have experienced a myocardial infarction (STEMI) within the previous 24 hours confirmed by symptoms and ECG.

Exclusion Criteria:

* Subjects with a known low ejection fraction of less than 40% or any previous history of heart failure.
* Subjects treated with eplerenone or other aldosterone antagonists within the past 1 month.
* The subject has uncontrolled hypotension (SBP<90mmHg).
* Subjects with eGFR ≤30ml/min (based on admission serum creatinine and the MDRD formula) or serum creatinine ≥220µmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - Walter C Mackenzie Health Sciences Centre (WCM), Edmonton, Alberta
  - Diamond Health Care Centre (DHCC), Vancouver, British Columbia
  - Vancouver General Hospital - Centennial Pavilion, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Health Sciences Center, Eastern Health, St. John's, Newfoundland and Labrador
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre de Sante et de Services Sociaux de Chicoutimi (CSSSC) (Complexe Hospitalier de la Sagamie), Chicoutimi, Quebec
  - ECOGENE-21 / Centre de sante et de services sociaux de Chicoutimi, Chicoutimi, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Hopital Fleurimont, Sherbrooke, Quebec
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - I.Interni klinika-kardiologie FN Olomouc, Olomouc
  - I. Interni klinika - kardiologie FN Olomouc, Olomouc
  - Klinika kardiologie IKEM, Prague
  - Nemocnice Na Homolce - kardiologicke oddeleni, Prague
- France (9):
  - Chu Rangueil Service de Cardiologie, A - Bat H1, Toulouse, Cedex 4
  - Chu du Bocage - Centre de Cardiologie, Dijon, Cedex
  - Hopital De La Pitie Salpetriere, Paris, Cedex
  - Service Cardiologie, Centre Hospitalier de Cannes, Cannes
  - Hôpital Henri Mondor - Pysiologie explorations fonctionnelles, Créteil
  - Hôpital Henri Mondor, Créteil
  - Centre de Cardiologie d'Evecquemont, Évecquemont
  - Service Cardiologie Hopital Robert Boulin, Libourne
  - Cardiologie Interventionnelle, Pessac
- Germany (13):
  - Universitaets-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Links der Weser gGmbH, Bremen
  - Sankt Johannes Hospital Medizinische Klinik I, Dortmund
  - Sankt Johannes Hospital, Dortmund
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Georg-August-Universitaet Goettingen, Zentrum f. Innere Medizin / Kardiologie u. Pneumologie, Göttingen
  - Universitaeres Herzzentrum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - St. Vincenz Krankenhaus, Limburg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Staedtisches Klinikum Muenchen GmbH Klinikum Neuperlach, Munich
- Greece (3):
  - General Hospital of Athens "Georgios Gennimatas", Athens
  - General Hospital of Attiki KAT, Athens
  - University General Hospital of Patra, Rio Patra
- Hungary (4):
  - Budai Irgalmasrendi Korhaz, Kardiologia, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Kardiologiai Osztaly, Győr
  - Josa Andras Oktato Korhaz Egeszsegugyi Szolgaltato Nonprofit Kft., Kardiologia, Nyíregyháza
  - Zala Megyei Korhaz, Kardiologia, Zalaegerszeg
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Locatie Oosterpark, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
- Poland (4):
  - Katedra i Klinika Kardiologii i Chorob Wewnetrznych, Bydgoszcz
  - Oddzial Kardiologiczny Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii NZOZ w Oswiecimiu G.V.M CARINT Sp. zo.o., Oświęcim
  - Oddzial Kardiologiczny Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw
- Slovakia (5):
  - Stredoslovensky ustav srdcovych a cievnych chorob, a.s., Banská Bystrica
  - Narodny ustav srdcovych a cievnych chorob, a.s., Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Kardiocentrum Nitra, s.r.o., Nitra
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
- Spain (7):
  - Hospital Del Sas de Jerez de La Frontera, Jerez de la Frontera, Cadiz
  - "Hospital Clinic i Provincial de Barcelona,Instituto Clinic del Torax, Barcelona
  - Hospital del Mar., Barcelona
  - HOSPITAL CLINICO SAN CARLOS- Universidad Complutense de Madrid, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (10):
  - Blackpool Victoria Hospital NHS Trust , Cardiac Research ,Lancashire Cardiac Centre, Blackpool, Lancashire
  - Edinburgh Royal Infirmary, Edinburgh, Lothian
  - Clinical Trials Unit Morriston Hospital, Swansea, Wales
  - City Hospital, Birmingham
  - Academic cardiology Unit, Cottingham Hull
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Ninewells Hospital and Medical School, Dundee
  - The Queens Medical Research Institute- University of Edinburgh, Edinburgh
  - University Hospital of Leicester (UHL) NHS Trust, Leicester
  - Clinical Trials Unit, Morriston Hospital, Swansea

REFERENCES:
- [Derived] Montalescot G, Pitt B, Lopez de Sa E, Hamm CW, Flather M, Verheugt F, Shi H, Turgonyi E, Orri M, Vincent J, Zannad F; REMINDER Investigators; REMINDER Investigators. Early eplerenone treatment in patients with acute ST-elevation myocardial infarction without heart failure: the Randomized Double-Blind Reminder Study. Eur Heart J. 2014 Sep 7;35(34):2295-302. doi: 10.1093/eurheartj/ehu164. Epub 2014 Apr 29. PMID 24780614
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141116&StudyName=Impact%20Of%20Eplerenone%20On%20Cardiovascular%20Outcomes%20In%20Patients%20Post%20Myocardial%20Infarction

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1012 subjects were enrolled for participation in this study. A total of 505 subjects were randomized to treatment with eplerenone and 505 subjects were randomized to the placebo group; a total of 422 and 424 subjects in the eplerenone and placebo groups, respectively, completed the study.
Groups:
- Eplerenone Plus Standard of Care: Eplerenone group received eplerenone 25 milligram (mg) once daily (OD), and on day 2, the dose of study drug increased to 50 mg OD (2 tablets) if serum potassium <5.0 mmol/L and with normal renal function.
- Placebo Plus Standard of Care: Placebo group received matching placebo for eplerenone 25 milligram (mg) film coated tablets.
Period: Overall Study
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Started | 506 | 506
Treated | 505 | 505
Completed | 422 | 424
Not Completed | 84 | 82
Not completed — Adverse Event | 10 | 11
Not completed — Death | 2 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 16 | 14
Not completed — Withdrawal by Subject | 48 | 48
Not completed — Protocol Violation | 2 | 1
Not completed — Did Not Meet Entrance Criteria | 1 | 0
Not completed — Study terminated by sponsor | 0 | 1
Not completed — Reason not defined | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care | Total
Number analyzed (Participants) | 506 | 506 | 1012
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (10.8) | 57.8 (11.0) | 58.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 103 | 189
  Male | 420 | 403 | 823

OUTCOME MEASURES:

1. Primary Outcome: First Event of Cardiovascular Mortality, Re-hospitalization or Extended Initial Hospital Stay Due to Diagnosis of Heart Failure, Sustained Ventricular Tachycardia or Fibrillation, Ejection Fraction ≤40% or BNP Above Age Adjusted Cut Off
Description: Cardiovascular mortality is defined as any mortality adjudicated as death due to sudden cardiac death, myocardial infarction (MI), worsening heart failure, cardiac arrhythmia, other cause (such as pulmonary embolism, peripheral arterial disease [PAD], etc.). Hospitalization due to congestive heart failure (CHF) and requires extended hospital stay or frequent visits to emergency room, observation unit or in-patient care, due to CHF as the primary or secondary diagnosis supported by a discharge report or clinical summary for hospitalization as determined by the endpoint adjudication committee (EAC). A composite of time to first event of cardiovascular mortality (CV), re-hospitalization or extended initial hospital stay due to diagnosis of heart failure, sustained ventricular tachycardia or fibrillation, ejection fraction ≤40% after 1 month or BNP >200 pg/mL or NT-proBNP >450 pg/mL (age <50 years); >900 pg/mL (age 50 to 75 years) or >1800 pg/mL (age >75 years) after 1 month.
Time Frame: 0-24 months
Population: The Full Analysis Set (FAS) using the intent-to-treat (ITT) principle, regardless of compliance with the study drug and the protocol was used. The efficacy analysis data sets for clinical events included all available study endpoints.
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 92 | 149
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; Hazard ratio, 95% confidence interval (CI) of hazard ratio, and p-value for the Primary Analysis based on a Cox proportional hazard model with treatment as the major factor, adjusted for baseline estimated glomerular filtration rate (eGFR), with/without previous MI, time of first dose administered post onset of index symptom, and location of index MI anterior or non-anterior; Test type: Superiority or Other; p < 0.0001, Regression, Cox — All analyses for primary endpoint were tested at two-sided, α-level of 0.05, without adjusting for multiplicity; Cox Proportional Hazard = 0.581, 95% CI 2-sided [0.446 to 0.756]

2. Secondary Outcome: Cardiovascular Mortality
Description: The occurrence of cardiovascular mortality from randomization. Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used. The efficacy analysis data sets for clinical events included all available study endpoints. Furthermore, only events confirmed by the EAC were used.
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 2 | 2
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; Hazard ratio, 95% CI of hazard ratio, p-value for all secondary endpoints based on Cox proportional hazard model with treatment as the major factor, adjusted for baseline eGFR, with/without previous MI, index MI location, time of first dose administered post onset of index symptom; Test type: Superiority or Other; p = 0.6406, Regression, Cox; Cox Proportional Hazard = 0.562, 95% CI 2-sided [0.050 to 6.308]

3. Secondary Outcome: Diagnosis of Heart Failure
Description: The occurrence of first diagnosis of heart failure from the date of randomization. Time-to-event analyses were measured from the date of randomization, and a subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: as for outcome 2
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 7 | 11
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; Hazard ratio, 95% CI of hazard ratio, p-value for all secondary endpoints based on Cox proportional hazard model with treatment as a factor, adjusted for baseline eGFR, with/without previous MI, index MI location, time of first dose administered post onset of index symptom; Test type: Superiority or Other; p = 0.5338, Regression, Cox; Cox Proportional Hazard = 0.726, 95% CI 2-sided [0.265 to 1.990]

4. Secondary Outcome: First and Each Subsequent Episode (After an Event Free Interval of ≥ 48 Hours) of Sustained Ventricular Tachycardia or Ventricular Fibrillation.
Description: The occurrence of first and each subsequent episode (after an event-free interval of ≥ 48 hours) of sustained ventricular tachycardia or ventricular fibrillation. Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: as for outcome 2
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 0 | 0

5. Secondary Outcome: First Recorded Ejection Fraction (EF) of ≤40% (Recorded 1 Month or Later Post-randomization).
Description: The occurrence of first recorded EF ≤40% (recorded 28 days or later post-randomization). Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used. The efficacy analysis data sets for clinical events included all available study endpoints.
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 20 | 19
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8042, Regression, Cox; Cox Proportional Hazard = 1.083, 95% CI 2-sided [0.575 to 2.040]

6. Secondary Outcome: Brain (B-type) Natriuretic Peptide (BNP) >200 pg/mL or NT-proBNP >450, >900 or >1800 pg/mL for Ages <50 Years, 50-75 Years and >75 Years, Respectively (Recorded 1 Month or Later Post-randomization).
Description: The occurrence of first occurrence of BNP >200 pg/mL or NT-proBNP >450, >900 or >1800 pg/mL for ages <50 years, 50 to 75 years and >75 years, respectively (recorded 28 days or later post-randomization). Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used.
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 81 | 131
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0003, Regression, Cox; Cox Proportional Hazard = 0.598, 95% CI 2-sided [0.452 to 0.791]

7. Secondary Outcome: Decision to Provide an Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy (CRT).
Description: The decision to provide an ICD or CRT. Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used.
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 3 | 3
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9353, Regression, Cox; Cox Proportional Hazard = 1.069, 95% CI 2-sided [0.213 to 5.371]

8. Secondary Outcome: Second or Subsequent Non-fatal Myocardial Infarction (MI).
Description: The occurrence of second or subsequent nonfatal MI. Time-to-event analyses were measured from the date of randomization. A subject who did not experience the endpoint(s) of interest was censored on the last day the subject was confirmed by the investigator to be endpoint-free. The time-to-event distributions were summarized by treatment group using Kaplan-Meier estimates of cumulative incidence.
Time Frame: 0-24 months
Population: as for outcome 2
Measure: Number; unit: Events
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Events | 10 | 6
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3757, Regression, Cox; Cox Proportional Hazard = 1.600, 95% CI 2-sided [0.566 to 4.525]

9. Secondary Outcome: Electrocardiogram Q Wave to the End of the S Wave Corresponding to Ventricle Depolarization (QRS) Duration at 6 Months Post-randomization.
Description: Electrocardiogram Q wave to the end of the S wave corresponding to ventricle depolarization (QRS) duration at 6 months post-randomization. The continuous endpoints were assessed using analysis of covariance (ANCOVA) model, fitted with corresponding baseline and treatment. These were analyzed at 6 months based on last observation carried forward (LOCF) and also using all available data up to end of study.
Time Frame: 6 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 347 | 343
Milliseconds (msec) | 93.31 (15.04) | 94.62 (16.00)
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; ANCOVA model was used with observed value as the dependent variable, treatment as a major factor, and baseline QRS duration, baseline eGFR, with/without previous MI, time (in hours) of first dose administered post onset of index symptom, and location of index MI (anterior versus all other locations) as covariates; Test type: Superiority or Other; p = 0.1744, ANCOVA; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-3.55 to 0.65]

10. Secondary Outcome: Left Atrial Diameter (LAD) (Recorded on Each Occasion an Echocardiogram is Conducted).
Description: LAD recorded each time an echocardiogram is conducted. The continuous endpoints were assessed using ANCOVA model, fitted with corresponding baseline and treatment. These were analyzed at 6 months based on LOCF and also using all available data up to end of study.
Time Frame: 0-24 months
Population: The FAS using the ITT principle, regardless of compliance with the study drug and the protocol was used.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 506 | 506
Centimeters (cm)
  Month 6 (N = 268, 243) | 3.92 (0.654) | 3.90 (0.703)
  Final Visit (N = 393, 378) | 3.91 (0.641) | 3.87 (0.658)
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For the Between-Treatment difference for Eplerenone and Placebo groups of observed value taken at Month 6 visit, ANCOVA model was performed for LAD based on the LOCF method including treatment groups with/without adjustments for baseline eGFR (in mL/min/1.73 m2), previous MI (yes/no), time (in hours) of first dose administered post-onset of symptom, index MI location (anterior versus all others) as covariates; Test type: Superiority or Other; p = 0.7123, ANCOVA — ANCOVA was used for between-treatment comparisons of the LSMeans, 95% CI of LSMEANS, LSMeans difference, 95% CI of LSMeans difference, and p-value with observed value at the given time point as variable; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.10 to 0.14]
Statistical Analysis 2: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.4105, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.05 to 0.13]

11. Secondary Outcome: Change in Serum Levels of Biomarkers (Aldosterone and Cortisol) at 6 Months Post-randomization.
Description: Change in serum levels of aldosterone and cortisol at 6 months post-randomization. The continuous endpoints were assessed using ANCOVA model, fitted with corresponding baseline and treatment. These were analyzed at 6 months based on LOCF and also using all available data up to end of study.
Time Frame: 6 months
Population: The Biomarker Analysis Set is a subset of FAS subjects who have the biomarker data (carboxyterminal telopeptide of type I collagen [ICTP], procollagen type I N-terminal peptide [PINP], procollagen type III N-terminal peptide [PIIINP], Interleukin-6, aldosterone, cortisol, and Galactin 3) available.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 266 | 260
nmol/L
  Aldosterone | 0.355 [0.210 to 0.540] | 0.210 [0.150 to 0.310]
  Serum Cortisol | 379.0 [292.0 to 492.0] | 366.0 [271.0 to 482.0]
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care; For Biomarker- Aldosterone, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 2: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p < 0.5552, Signed Rank Test
Statistical Analysis 3: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- Aldosterone, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank-Sum test
Statistical Analysis 4: Comparison: Eplerenone Plus Standard of Care; For Biomarker- Serum Cortisol, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 5: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 6: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- Serum Cortisol, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.3347, Wilcoxon Rank-Sum test

12. Secondary Outcome: Change in Serum Levels of Biomarkers (PIIINP, Galectin 3, and PINP) at 6 Months Post-randomization.
Description: Change in serum levels of PIIINP, Galectin 3, and PINP at 6 months post-randomization. The continuous endpoints were assessed using ANCOVA model, fitted with corresponding baseline and treatment. These were analyzed at 6 months based on LOCF and also using all available data up to end of study.
Time Frame: 6 months
Population: The Biomarker Analysis Set is a subset of FAS subjects who have the biomarker data (ICTP, PINP, PIIINP, Interleukin-6, aldosterone, cortisol, and Galactin 3) available.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 266 | 260
ng/mL
  PIIINP | 4.20 [3.50 to 4.90] | 4.30 [3.60 to 5.10]
  Galectin 3 | 11.20 [9.20 to 13.50] | 10.60 [9.10 to 12.40]
  PINP | 30.0 [24.0 to 39.0] | 32.0 [24.0 to 42.0]
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care; For Biomarker- PIIINP, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p = 0.0005, Signed Rank Test
Statistical Analysis 2: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 3: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- PIIINP, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.1558, Wilcoxon-Rank Sum test
Statistical Analysis 4: Comparison: Eplerenone Plus Standard of Care; For Biomarker- Galecting 3, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p = 0.0008, Signed Rank Test
Statistical Analysis 5: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 6: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- Galecting 3, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.0293, Wilcoxon Rank-Sum test
Statistical Analysis 7: Comparison: Eplerenone Plus Standard of Care; For Biomarker- PINP, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p = 0.1723, Signed Rank Test
Statistical Analysis 8: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.0295, Signed Rank Test
Statistical Analysis 9: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- PINP, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.0865, Wilcoxon Rank-Sum test

13. Secondary Outcome: Change in Serum Level of Biomarker (ICTP) at 6 Months Post-randomization.
Description: Change in serum level of ICTP at 6 months post-randomization. The continuous endpoint was assessed using ANCOVA model, fitted with corresponding baseline and treatment. It was analyzed at 6 months based on LOCF and also using all available data up to end of study.
Time Frame: 6 months
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: μg/L
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 266 | 260
μg/L | 3.70 [3.20 to 4.50] | 3.70 [3.20 to 4.80]
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care; For Biomarker- ICTP, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p = 0.0944, Signed Rank Test
Statistical Analysis 2: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0360, Signed Rank Test
Statistical Analysis 3: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- ICTP, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.6459, Wilcoxon Rank-Sum test

14. Secondary Outcome: Change in Serum Level of Biomarker (Interleukin-6) at 6 Months Post-randomization.
Description: Change in serum level of Interleukin-6 at 6 months post-randomization. The continuous endpoint was assessed using ANCOVA model, fitted with corresponding baseline and treatment. It was analyzed at 6 months based on LOCF and also using all available data up to end of study.
Time Frame: 6 months
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 266 | 260
pg/mL | 1.845 [1.235 to 2.955] | 1.755 [1.180 to 2.480]
Statistical Analysis 1: Comparison: Eplerenone Plus Standard of Care; For Biomarker- Interleukin-6, signed rank test for change from baseline at Month 6 within treatment difference was used to derive p-value; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 2: Comparison: Placebo Plus Standard of Care; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Signed Rank Test
Statistical Analysis 3: Comparison: Eplerenone Plus Standard of Care vs Placebo Plus Standard of Care; For Biomarker- Interleukin-6, Wilconxon rank-sum test for between treatment difference at Month 6 was used to derive p-value; Test type: Superiority or Other; p = 0.0801, Wilcoxon Rank-Sum test

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Eplerenone Plus Standard of Care | Placebo Plus Standard of Care
Serious Adverse Events (participants affected / at risk) | 100/505 | 101/505
Other Adverse Events (participants affected / at risk) | 151/506 | 153/506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone Plus Standard of Care (N=505) | Placebo Plus Standard of Care (N=505)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 4
Angina pectoris (Cardiac disorders) | 12 | 10
Angina unstable (Cardiac disorders) | 4 | 9
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 9
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 4
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 2
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Long QT syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 2 | 0
Pericardial disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 3 | 2
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 4 | 9
Death (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 2
Sudden death (General disorders) | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0 — Device related infection
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Lung squamous cell carcinoma stage unspecified
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral artery thrombosis (Nervous system disorders) | 0 | 1 — Cerebral artery thrombosis
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Multiple system atrophy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 3 | 4
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 — Urinary bladder haemorrhage
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Chronic obstructive pulmonary disease
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Idiopathic pulmonary fibrosis
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 1 — Implantable defibrillator insertion
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0 — Inguinal hernia repair
Percutaneous coronary intervention (Surgical and medical procedures) | 1 | 0 — Percutaneous coronary intervention
Circulatory collapse (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1
Ischaemia (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 2 — Peripheral arterial occlusive disease
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone Plus Standard of Care (N=506) | Placebo Plus Standard of Care (N=506)
Angina pectoris (Cardiac disorders) | 16 | 22
Bradycardia (Cardiac disorders) | 12 | 7
Ventricular tachycardia (Cardiac disorders) | 11 | 7
Abdominal pain upper (Gastrointestinal disorders) | 13 | 3
Constipation (Gastrointestinal disorders) | 7 | 13
Diarrhoea (Gastrointestinal disorders) | 22 | 14
Nausea (Gastrointestinal disorders) | 7 | 11
Chest pain (General disorders) | 23 | 24
Fatigue (General disorders) | 10 | 20
Non-cardiac chest pain (General disorders) | 16 | 13
Oedema peripheral (General disorders) | 8 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 13
Dizziness (Nervous system disorders) | 21 | 19
Headache (Nervous system disorders) | 8 | 16
Anxiety (Psychiatric disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 17
Hypertension (Vascular disorders) | 12 | 18
Hypotension (Vascular disorders) | 21 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.